CLINICAL TRIAL: NCT00475683
Title: Randomized Cross-over Study of Curcumin for Prevention of Oral Mucositis in Children Receiving Doxorubicin Based Chemotherapy.
Brief Title: Curcumin for Prevention of Oral Mucositis in Children Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Shoshana Vilk, Prof. Shoshana Revel-Villk, Hadassah Medical Organization
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Curcumin-HMO-CTIL
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2011-06

CONDITIONS: Chemotherapy Induced Mucositis
Keywords: Doxorubicin; Mucositis; Prevention; Curcumin
MeSH Terms: conditions — Mucositis | interventions — Mouthwashes; curcumol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- regular measurments (Sham Comparator): Mouth wash with chlorexidin
  Interventions: Other: Mouth wash
- Curucmol (Experimental): mouth wash with curcumol and mouth wash with chlorexidin
  Interventions: Dietary Supplement: Curcumol

INTERVENTIONS:
Other: Mouth wash — Mouth wash with chlorehexidin, three times a day
  Arms: regular measurments
Dietary Supplement: Curcumol — 5 ml in 50 ml water, mouthwash for 30 seconds, three times a day
  Arms: Curucmol

SUMMARY:
Mucositis consists of inflammation of the mucosal membrane and is a prominent cause of patient discomfort during cancer therapy. In children receiving chemotherapy, the incidence of oral mucositis is reported to be between 40%-70%. Curcumin, a commonly-used spice in India and Southeast Asia, was shown in animal models to prevent chemotherapy and radiotherapy induced mucositis. We hypothesize that curcumin may prevent oral mucosal injury and reduce the severity of oral mucositis in children receiving chemotherapy. Thus, the aim of this study is to determine whether in children undergoing doxorubicin-containing chemotherapy, does supplementation of curcumin, when compared to placebo, decrease oral mucositis both by objective (mucositis scales) and subjective (pain scale) measurements. Effective prevention and reduction of mucosal injury may significantly improve the care we provide to children undergoing therapy for cancer.

DETAILED DESCRIPTION:
Children older than 5 years of age diagnosed with cancer and treated at the Pediatric Hematology/Oncology unit, Hadassah Medical Center will be eligible to the study. The study is designed as a cross-over study, wherein each patient serves as his or her own control, thus all included children should be scheduled to receive at least two identical curses of doxorubicin-containing chemotherapy in which the dose of doxorubicin is at least 60mg/m2 per course. The patients will be assigned to randomly receive curcumin or placebo in the 1st course, with the other regimen administered at the 2nd course. Curcumin will be given as fluid extract (1:1) at a dose of 10 drops, three times a day. Adolescents and young adults will receive the adult recommend dose, i.e. 30 drops, three times a day. Placebo will be given at the same dose. The patients will be taught to rinse the mouth with the medicine and than spit out. The therapy will be given from a day prior to the first day of the cycle for two weeks. A diary kept by the family will record each given dose. Possible side effects associated with the study drug, such as vomiting, nausea, rash, etc., will be recorded. No other adjunctive topical treatment will be used during the study. Adherence will be assessed through subject reports as well as by review of returned medications every cycle collected during the objective assessment site visits. Given the intent-to-treat analysis, all participants will be included irrespective of how much of the study medication was taken.The measurements of study outcome, i.e. OMAS score, WHO mucositis scale and visual analogue pain scale will be done on day 1,7,10,14,21 ± 1 of each chemotherapy cycle. The following data will be recorded in all cycles: duration of neutropenia, the need and length of hospitalization, use and dosage of opioid analgesia, need for total potential nutrition, blood culture positive infection and other mucositis related complications.

ELIGIBILITY:
Inclusion Criteria:

1. Children older than 5 years of age, adolescents and young adults diagnosed with cancer and treated at the Pediatric Hematology/Oncology unit, Hadassah Medical Center,
2. A crossover study design is planed wherein each patient serves as his or her own control, thus all included children should be scheduled to receive at least two identical curses of doxorubicin-containing chemotherapy in which the dose of doxorubicin is at least 60mg/m2 per course,
3. Patient's/ parent's informed consent.

Exclusion Criteria:

1. Patients treated with antiplatelet therapy or anticoagulation,
2. Patients with biliary tract obstruction,
3. Patients with preexisting oral disease, such as active oral infection, trauma to the oral mucosa or oral ulceration prior to chemotherapy,
4. Patients receiving head and neck radiation,
5. Developmentally unable to comply with curcumin mouth wash as judged by the parent or investigator.

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To determine whether in children undergoing doxorubicin-containing chemotherapy, does supplementation of curcumin, when compared to placebo, decrease an objective measurement of oral mucositis? | 6 weeks

SECONDARY OUTCOMES:
To determine whether in children undergoing doxorubicin-containing chemotherapy, does supplementation of curcumin, when compared to placebo, decrease mucositis related pain, use of opioids and parenteral nutrition. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shoshana Revel-Vilk, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel